CLINICAL TRIAL: NCT02455388
Title: d13C Added Sugar Intake Biomarker: Determining Validity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Hawaii (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Brenda Davy, Associate Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21HD078636-01A1 (NIH); R21HD078636 (NIH)
Record Dates: First submitted 2015-05-18; First posted 2015-05-27 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Validation Studies
Keywords: Nutrition; Obesity; Pediatric
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Study 1: Crossover design Study 2: Cross-sectional design
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low, then high added sugar diet (Experimental): Participants will consume a low added sugar (5% total energy) diet for 7 consecutive days. After a 4-week washout period, participants will then consume a high added sugar (25% total energy) diet for 7 consecutive days.
  Interventions: Dietary Supplement: High added sugar diet; Dietary Supplement: Low added sugar diet
- High, then low added sugar diet (Experimental): Participants will consume a high added sugar (25% total energy) diet for 7 consecutive days. After a 4-week washout period, participants will then consume a low added sugar (5% total energy) diet for 7 consecutive days
  Interventions: Dietary Supplement: High added sugar diet; Dietary Supplement: Low added sugar diet
- Dietary recall and fingerstick (No Intervention): Participants will complete 4 in-person 24-hr dietary recalls and 2 fingerstick blood samples at Visit 1 and 3 within 3 weeks.

INTERVENTIONS:
Dietary Supplement: High added sugar diet — Controlled feeding study. Participants will be provided with daily coolers containing foods with high (25%) added sugar to consume for 7 consecutive days. Fasting fingerstick blood samples and weight checks will be performed each morning.
  Arms: High, then low added sugar diet; Low, then high added sugar diet
Dietary Supplement: Low added sugar diet — Controlled feeding study. Participants will be provided with daily coolers containing foods with low (5%) added sugar to consume for 7 consecutive days. Fasting fingerstick blood samples and weight checks will be performed each morning.
  Arms: High, then low added sugar diet; Low, then high added sugar diet

SUMMARY:
Added sugars (AS) constitute a significant source (~ 16%) of the total daily calories consumed by youth. The role of AS in health is contentious, and the reliance on self-reported dietary data is an often-cited flaw in existing research. The investigators propose to establish the validity of the d13C biomarker for AS intake from fingerstick blood samples in children; our findings could significantly advance research addressing the health impacts of AS intake in children and adolescents.

DETAILED DESCRIPTION:
Consumption of energy-containing added sugars (AS) and in particular, sugar-sweetened beverages (SSB), have been suggested as contributors to weight gain. In children and adolescents, total AS intake represents ~16% of total energy, or ~300-400 kcal/d; SSB comprise ~50% of total AS intake. Although recognized by major health organizations, the role of AS and their primary food source, SSB, in the development and progression of obesity and related co-morbidities remains controversial. A common research limitation in this area is a reliance on self-reported measures of dietary intake, which present additional challenges when studying children. Thus, the need for objective methods to assess dietary intake, such as biomarkers of AS consumption, has been recognized. The investigators have established the validity of the fingerstick blood d13C AS biomarker in adults, and aim to expand our innovative biomarker to studies of diet in children. The investigators propose to establish the validity and reliability of the fingerstick blood d13C AS biomarker in children using two approaches. First, a controlled feeding component (Study 1) will provide data necessary for validation of the biomarker with actual AS intake, and determine its ability to detect levels of AS intake. Second, a cross-sectional component (Study 2) will compare the biomarker to self-reported intake data, collected in a method similar to national nutritional surveillance methodology (i.e., NHANES). Study 1 will include 30 adolescents aged 12-18 yrs, who will consume both a high AS (25% total energy) and low AS (5% total energy) diet for 7 days each, in a random order. Study 2 will include 325 children aged 6-18 yrs, who will complete five laboratory sessions. Record- assisted 24-hr dietary recalls will be completed at four of the sessions to assess habitual AS intake, and fingerstick blood samples will be obtained at two of the sessions. The potential confounding effects of non- sweetener corn and animal product consumption will be addressed in both studies by quantifying non- sweetener corn consumption in the controlled diets (Study 1) and in self-reported dietary recalls (Study 2), and by assessing the nitrogen stable isotope composition d15N of fingerstick samples. To advance existing knowledge of dietary assessment approaches, urinary sugars and urine d13C will be assessed in Study 1, which will permit a direct comparison of biomarkers - existing (urinary sucrose, fructose) and novel (urine and fingerstick d13C ). The role of AS in health has been contentious for decades, and the reliance on self-reported intake data is an often-cited flaw in this area. Our findings could significantly advance research addressing the health impacts of AS intake in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Cross-sectional study: Age 6-18, both genders
* Controlled feeding study: Age 12-18, both genders, BMI <95%ile

Exclusion Criteria:

* Controlled feeding study: Food allergies and/or aversions, BMI>95%ile

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 370 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda M Davy, Ph.D., Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States

REFERENCES:
- [Derived] MacDougall CR, Hill CE, Jahren AH, Savla J, Riebl SK, Hedrick VE, Raynor HA, Dunsmore JC, Frisard MI, Davy BM. The delta13C Value of Fingerstick Blood Is a Valid, Reliable, and Sensitive Biomarker of Sugar-Sweetened Beverage Intake in Children and Adolescents. J Nutr. 2018 Jan 1;148(1):147-152. doi: 10.1093/jn/nxx017. PMID 29378049
- [Derived] Moore LB, Liu SV, Halliday TM, Neilson AP, Hedrick VE, Davy BM. Urinary Excretion of Sodium, Nitrogen, and Sugar Amounts Are Valid Biomarkers of Dietary Sodium, Protein, and High Sugar Intake in Nonobese Adolescents. J Nutr. 2017 Dec;147(12):2364-2373. doi: 10.3945/jn.117.256875. Epub 2017 Sep 20. PMID 28931586

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events took place in the study after enrollment but prior to arm assignment.
Groups:
- Low, Then High Added Sugar Diet: Participants will consume a low added sugar (5% total energy) diet for 7 consecutive days. After a 4-week washout period, participants will consume a high added sugar (25% total energy) diet for 7 consecutive days.
  Low and high added sugar diet: Controlled feeding study. Participants will be provided with daily coolers containing foods with low (5%) or high (25%) added sugar to consume for 7 consecutive days. Fasting fingerstick blood samples and weight checks will be performed each morning.
- High, Then Low Added Sugar Diet: Participants will consume high added sugar (25% total energy) diet for 7 consecutive days. After a 4-week washout period, participants will consume a low added sugar (5% total energy) diet for 7 consecutive days.
  High and low added sugar diet: Controlled feeding study. Participants will be provided with daily coolers containing foods with high (25%) or low (5%) added sugar to consume for 7 consecutive days. Fasting fingerstick blood samples and weight checks will be performed each morning.
- Dietary Recall and Fingerstick: Participants will complete 4 in-person 24-hr dietary recalls and 2 fingerstick blood samples at visits 1 and 3 within 3 weeks.
Period: Overall Study
Arm/Group | Low, Then High Added Sugar Diet | High, Then Low Added Sugar Diet | Dietary Recall and Fingerstick
Started | 18 | 15 | 337
Completed | 17 | 15 | 326
Not Completed | 1 | 0 | 11
Not completed — Protocol Violation | 1 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: The baseline analysis population does not include 11 individuals who either voluntarily withdrew from the study or did not provide all fingerstick blood samples (Cross-sectional study).
Groups:
- Controlled Feeding Study: Participants will be randomly assigned to consume either a high (25% total energy) or low (5% total energy) added sugar diet for the first 7 consecutive day period. After a 4-week washout period, participants will then consume the other diet for another period of 7 consecutive days.
  High added sugar diet: Controlled feeding study. Participants will be provided with daily coolers containing foods with high (25%) added sugar to consume for 7 consecutive days. Fasting fingerstick blood samples and weight checks will be performed each morning.
  Low added sugar diet: Controlled feeding study. Participants will be provided with daily coolers containing foods with low (5%) added sugar to consume for 7 consecutive days. Fasting fingerstick blood samples and weight checks will be performed each morning.
- Cross-sectional Study: Participants will complete 4 in-person 24-hr dietary recalls within 3 weeks and 2 fingerstick blood samples at Visit 1 and 3.
- Total: Total of all reporting groups
Arm/Group | Controlled Feeding Study | Cross-sectional Study | Total
Number analyzed (Participants) | 32 | 326 | 358
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 326 | 358
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.6) | 12 (3) | 12.6 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 167 | 184
  Male | 15 | 159 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 6 | 6
  Not Hispanic or Latino | 31 | 303 | 334
  Unknown or Not Reported | 1 | 17 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 7 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 32 | 313 | 345
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 32 | 326 | 358
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 20.2 (2.1) | 20.0 (4.5) | 20.0 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: delta13C Added Sugar Biomarker
Description: Validity, reliability, and sensitivity of the fingerstick blood d13C AS biomarker during cross-sectional data collection. Participants will provide 4 separate self-reported, record-assisted 24-hr food intake recalls, and at two of the visits, a fingerstick blood sample will be collected to analyze delta13C biomarker levels.
Time Frame: 2-3 weeks
Measure: Mean (Standard Deviation); unit: ‰ δ13C
Arm/Group | Cross-sectional Study
Number analyzed (Participants) | 326
‰ δ13C
  Visit 1 | -19.66 (0.68)
  Visit 3 | -19.64 (0.68)
Statistical Analysis 1: Comparison: Cross-sectional Study; Test type: Equivalence — No equivalence margin set; p < 0.001, Intraclass correlation coefficient

2. Secondary Outcome: Change in d13C: delta13C Added Sugar Biomarker
Description: Validity, reliability and sensitivity of the fingerstick blood delta13C AS biomarker during feeding study. Participants are provided 7 days of food with high or low added sugar diet. Blood samples will be obtained each day via fingerstick to analyze delta13C biomarker levels.
Time Frame: Two 7-day feeding periods, randomized order, with a four-week washout between feeding periods. Outcome is a change in d13C from day 1 to 8, for each feeding period.
Population: Adolescents aged 12-18 years with a body mass index percentile <95%. They were willing to follow a controlled diet and did not have food allergies, intolerances or aversions.
Measure: Mean (Standard Deviation); unit: ‰
Groups:
- Low Added Sugar Diet: Participants will consume a low added sugar (5% total energy) diet for 7 consecutive days.
  Low and high added sugar diet: Controlled feeding study. Participants will be provided with daily coolers containing foods with low (5%) or high (25%) added sugar to consume for 7 consecutive days. Fasting fingerstick blood samples and weight checks will be performed each morning.
- High Added Sugar Diet: Participants will consume high added sugar (25% total energy) diet for 7 consecutive days.
  High and low added sugar diet: Controlled feeding study. Participants will be provided with daily coolers containing foods with high (25%) or low (5%) added sugar to consume for 7 consecutive days. Fasting fingerstick blood samples and weight checks will be performed each morning.
Arm/Group | Low Added Sugar Diet | High Added Sugar Diet
Number analyzed (Participants) | 32 | 32
‰ | -0.05 (0.071) | 0.03 (0.083)
Statistical Analysis 1: Comparison: Low Added Sugar Diet vs High Added Sugar Diet; Test type: Superiority; p < 0.05, ANOVA

3. Secondary Outcome: Diagnostic Value of d13C Biomarker
Description: Determine diagnostic value of d13C biomarker using fingerstick blood. The area under the ROC was used as a measure for the diagnostic accuracy of the d13C biomarker, with values closer to 1.0 indicating greater ability to distinguish between low and high added sugar and sugar sweetened beverage consumers.
Time Frame: 2-3 weeks
Measure: Number (95% Confidence Interval); unit: Area under the ROC curve
Arm/Group | Cross-sectional Study
Number analyzed (Participants) | 326
Area under the ROC curve | 0.61 [0.56 to 0.67]
Statistical Analysis 1: Comparison: Cross-sectional Study; Test type: Other; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 1.70

ADVERSE EVENTS:
Time Frame: 2.5 years
Groups:
- Cross-sectional Study: Participants will complete 4 in-person 24-hr dietary recalls and 2 fingerstick blood samples at Visit 1 and 3 within 3 weeks.
Arm/Group | Low, Then High Added Sugar Diet | High, Then Low Added Sugar Diet | Cross-sectional Study
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/337
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/337
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/337

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes